CLINICAL TRIAL: NCT05264051
Title: MAsS Scan as a Predictor of Morbidity and Mortality in Patients With Liver Disease
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB21-0900
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to study the muscle assessment score (MAsS, utilizing MRI, as an objective measure of frailty and muscle composition to serve as a predictor of morbidity and mortality in patients with liver disease.

DETAILED DESCRIPTION:
Prospective study of patients seen at the Univ. of Chicago Medical Center hospital and ambulatory clinics. The assessment of the MAsS score will require an additional 8-10 minutes in the MRI for each patient already undergoing MRI exam.

Four groups of pts. who are already scheduled for MRI for routine clinical purposes will be evaluated.

1. Pts. hospitalized with acute hepatic decompensation for whom MRI is otherwise indicated for clinical evaluation.
2. Pts. with hepatobiliary neoplasia
3. Pts.undergoing transjugular portosystemic shunt (TIPS) placement
4. Pts. with chronic liver disease undergoing magnetic resonance elastography for routine monitoring

ELIGIBILITY:
Inclusion Criteria:

* Patients who are already scheduled for an MRI for routine clinical purposes will be evaluated

Exclusion Criteria:

* <18 yrs. of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pts. hospitalized with acute hepatic decompensation Pts. with hepatobiliary neoplasia Pts. undergoing TIPS placement Pts. with chroinic liver disease
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Waitlist Mortality | Measured up to 10 years out from enrollment
  Death prior to liver transplant or delisting from enrollment in the study

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States